CLINICAL TRIAL: NCT03436680
Title: Feasibility of Home-Based Neurofeedback to Treat Chemotherapy-Induced Peripheral Neuropathy
Brief Title: Home-Based Neurofeedback Program in Treating Participants With Chemotherapy-Induced Peripheral Neuropathy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to lack of funds, time, and staff cannot activate the study.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2017-0309; NCI-2018-01049 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2017-0309 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2018-01-26; First posted 2018-02-19 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-02

CONDITIONS: Neuropathy
MeSH Terms: interventions — Practice Guidelines as Topic; Standard of Care; Neurofeedback

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (neurofeedback) (Experimental): Participants complete at least neurofeedback training sessions over 30 minutes 2 times a week for up to 5 weeks.
  Interventions: Other: Best Practice; Behavioral: Neurofeedback; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Group II (standard of care) (Active Comparator): Participants receive standard of care.
  Interventions: Other: Best Practice; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Other: Best Practice — Receive standard of care
  Other Names: standard of care; standard therapy
Behavioral: Neurofeedback — Complete neurofeedback training sessions
  Other Names: EEG biofeedback
  Arms: Group I (neurofeedback)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This trial studies how well a home-based neurofeedback program works in treating participants with chemotherapy-induced peripheral neuropathy (nerve damage that affects motor function). Neurofeedback training is a type of therapy that uses an electroencephalograph and a computer software program to measure brain wave activity. It may help teach participants how to change their own brain waves to lower their perception of pain symptoms and improve overall quality of life.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Examine the feasibility of using a home-based neurofeedback system and dry electroencephalography (EEG) cap to treat chemotherapy-induced peripheral neuropathy (CIPN).

SECONDARY OBJECTIVES:

I. Estimate the effects of home-based neurofeedback (HBNF) on symptoms of (CIPN) versus a wait list (WL) control group in cancer patients.

II. Estimate the effects of home-based neurofeedback (HBNF), versus WL, on the cortical and subcortical brain regions associated with CIPN.

III. Estimate the effects of a HBNF on other aspects of pain, cancer-related symptoms, quality of life (QOL), and mental health.

OUTLINE: Participants are randomized to 1 of 2 groups.

GROUP I: Participants complete at least neurofeedback training sessions over 30 minutes 2 times a week for up to 5 weeks.

GROUP II: Participants receive standard of care.

After completion of study, participants are followed up at 1 week for Group I and 6 weeks for Group II.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have the ability to understand and read English, sign a written informed consent, and be willing to follow protocol requirements.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
* Neuropathic pain score >= 4 on a 0-10 numeric pain scale (numeric rating scale [NRS]) and/or grade 3 or higher neuropathic symptoms according to the National Cancer Institute's 4 point grading scale.
* Neuropathic symptoms must be related to chemotherapy (in the opinion of the treating physician).
* Patients must have had neuropathic symptoms for a minimum of 3 months.
* No plans to change pain medication regimen during the course of the study.
* Off active chemotherapy treatment for minimum of 6 months.
* Hormonal (e.g., tamoxifen or arimidex, etc.) and targeted (tarceva and avastin, etc.) therapies allowed as long as they will be continued during the course of the study.
* Willing to come to MD Anderson for the intake and follow up data acquisition and to receive their equipment.
* Willing to allow research staff to come to their homes or to return the equipment to MD Anderson (MDA) in the case of equipment malfunction.
* Have had a diagnosis of cancer treated with chemotherapy.
* Live within a 50 mile radius of MD Anderson's main campus.

Exclusion Criteria:

* Patients who are taking any antipsychotic medications.
* Patients with active central nervous system (CNS) disease, such as clinically-evident metastases or leptomeningeal disease, dementia, or encephalopathy.
* Patients who have ever been diagnosed with bipolar disorder or schizophrenia.
* Patients with known, previously diagnosed peripheral neuropathy from causes other than chemotherapy.
* Patients who have a history of head injury or who have known seizure activity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of a Home-Based Neurofeedback (HBNF) System | 6 weeks
  HBNF intervention feasible if the average number of HBNF sessions completed across patients in the HBNF arm is >= 15.0 (or on average the proportion of sessions completed is >= 75%).

SECONDARY OUTCOMES:
Effects of Home-Based Neurofeedback (HBNF) on Symptoms of Chemotherapy-Induced Peripheral Neuropathy (CIPN) Versus a Waitlist (WL) Control Group in Cancer Patients | Baseline and at 6 weeks
  Summary statistics and 90% confidence intervals calculated for the Pain Quality Assessment Scale (PQAS) rated from 0 - 10 by study arm at baseline and at the end of treatment.
Effects of Neurofeedback on the Cortical and Subcortical Brain Regions Associated with Chemotherapy-Induced Peripheral Neuropathy (CIPN) and Effects of Home-Based Neurofeedback (HBNF) versus Waitlist (WL) Control Group determined by EEG, | Baseline and at 6 weeks
Effects of Home-Based Neurofeedback (HBNF) on Other Aspects of Cancer-Related Symptoms Using Patient Surveys | Baseline and within 7 days of the conclusion of treatment.
Effects of Home-Based Neurofeedback (HBNF) on Symptoms of Chemotherapy-Induced Peripheral Neuropathy (CIPN) Versus a Waitlist (WL) Control Group in Cancer Patients | Baseline and at 6 weeks
  Summary statistics and 90% confidence intervals calculated for the Brief Pain Inventory Short Form (BPI) by study arm at baseline and at the end of treatment.
Effects of Neurofeedback on the Cortical and Subcortical Brain Regions Associated with CIPN Determined by Changes in EEG as Measured by Low Resolution Electromagnetic Tomography (LORETA). | Baseline and at 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Prinsloo, Principal Investigator — M.D. Anderson Cancer Center

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org